CLINICAL TRIAL: NCT01527539
Title: A Multi-centre, Non-comparative, Open-labelled, Extension Trial to Assess the Long Term Safety and Efficacy of Biphasic Insulin Aspart 30 in Subjects With Type 2 Diabetes (Extension to BIAsp-1237)
Brief Title: Long Term Safety and Efficacy of Biphasic Insulin Aspart 30 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1479
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIAsp 30 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Dose individually adjusted. Injected twice daily immediately before breakfast and dinner. Administrated subcutaneously (s.c., under the skin)

SUMMARY:
This trial is conducted in North America. The aim of this trial is asses the long term safety and efficacy of biphasic insulin aspart 30 in Canadian subjects with type 2 diabetes who had participated in the BIAsp-1237 trial.

ELIGIBILITY:
Inclusion Criteria:

* Completed the BIAsp-1237 trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-11-23 (Actual); Primary Completion 2004-10-12 (Actual); Study Completion 2004-10-12 (Actual)

PRIMARY OUTCOMES:
HbA1c

SECONDARY OUTCOMES:
Occurrence of adverse events
Occurence of hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- Canada (4):
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Edmonton
  - Novo Nordisk Investigational Site, Windsor

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com